CLINICAL TRIAL: NCT06527274
Title: Effect of Defocus in Soft Contact Lenses on Internal Retinal Vascularization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2024-5133
Record Dates: First submitted 2024-07-08; First posted 2024-07-30 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Nearsightedness
Keywords: myopia; retinal vasculature; choroidal thickness
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, crossover masked study. Participants are randomly assigned to wear one type of soft lens for one week, then washed out for a few days, and then the second type of soft lens for the same period of time. Participants are masked to the type of lens provided
Who Masked: Participant
Masking Description: The lenses used in this study are daily disposable. This means that for each type of lens worn, participants will receive 7 lenses of each type. Lenses will be delivered one type at a time for the next week. The lenses will be packaged with a neutral label with a lot number. It is impossible for the participant to know which type this lot number corresponds to. Therefore, they do not know what type of lens they will receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myopic defocus soft lens design (MDSL) (Experimental): This arm involves the wear of a daily disposable soft contact lens (nesofilcon A) designed with a myopic defocus zone. This is a 14.2mm total diameter lens with a 4.2mm central zone for distance vision correction. This is followed by an abrupt transition zone of 1.2mm with no optical power. Then a higher convex power zone covers the surface to the edge of the optical zone (8mm). The rest of the lens (up to 14.2 mmOAD) supports the lens on the eye surface and has no power nor refractive effect. The power of the add area is calibrated to the central power to achieve a net add power of +5D. For example: -1.00D central power is surrounded by a +6D convex area; -2D is surrounded by a +7D area, and so on.)
  Interventions: Device: Experimental: Myopic defocus soft lens design (MDSL)
- Single vision soft lens design (SVSL) (Active Comparator): This arm involves the wear of a daily disposable soft contact lens (nesofilcon A) designed as a regular optical device to compensate for refractive error. In the case of this study, this lens will be made available from -1.00D to -4.00D. This lens is already in regular use in the US (K113703) and Canadian markets. Its design includes a central optical zone of 8mm that is powered to correct distance vision. The rest of the lens is supported on the ocular surface and has no power.
  Interventions: Device: Active Comparator: Single vision soft lens design (SVSL

INTERVENTIONS:
Device: Experimental: Myopic defocus soft lens design (MDSL) — An optical device designed to provide a myopic defocus to control myopia progression
  Arms: Myopic defocus soft lens design (MDSL)
Device: Active Comparator: Single vision soft lens design (SVSL — An optical device designed to correct refractive error like myopia
  Arms: Single vision soft lens design (SVSL)

SUMMARY:
The purpose of this study is to gain a better understanding of the retinal vascular changes that occur in response to the optical effect of a myopic defocus daily disposable soft contact lens (MDSL) in a group of healthy young myopic adults (18-35 years; myopia -1.00D to -4.00D; all genders). It will also learn about the acceptance of this visual correction modality compared to regular contact lenses.

The main questions to be answered are:

* To evaluate changes in retinal blood flow by visualizing retinal vascular density in the superficial and deep plexus after one week of MDSL wear.
* To evaluate changes in choroidal thickness at the macular level after one week of MDSL wear.
* To evaluate the visual comfort provided by this MDSL design using a questionnaire.

Researchers will compare the MDSL to a daily disposable single vision soft lens (SVSL) used to correct myopia to determine if the addition of a defocus area makes a difference in the retinal response to the visual signal.

Participants will be required to

* Wear both MDSL and SVSL for one week each, in a random order.
* Read letters to measure visual acuity
* Have a deep scan of their retina with an optical coherence tomography (OCT) device
* Rate the comfort and vision provided by both devices using a questionnaire.

DETAILED DESCRIPTION:
Objective:

The aim of this study is to gain a better understanding of the retinal vascular changes that occur in response to the optical effect of a myopic defocus daily disposable contact lens used in another (ongoing) research project (NCT05191134).

The primary objective of the study is to evaluate changes in retinal blood flow by visualizing retinal vascular density in the superficial and deep plexus following one week's wear of a high peripheral add soft contact lens in a population of young myopic adults.

The second objective is to assess changes in choroidal thickness at the macular level after one week's wear of the high peripheral add soft contact lens.

A third objective is to evaluate, through questionnaire, the visual comfort provided by this lens design.

Materials and methods:

25 myopic participants aged between 18 and 35 will be enrolled. Each participant will be randomly fitted with two lenses: a monofocal spherical soft lens (nesofilcon A) for one week and a high-add bifocal soft lens (anti-myopia) for the same duration of time. Participants will be asked to attend three different visits, one week apart.

At visit #1, initial measurements of deep and superficial plexus blood vessel density and choroidal thickness will be taken with an angiographic optical coherence tomograph (OCT-A Triton, Topcon USA).

These measurements will be repeated with other lenses at visit 2 and 3.

The results will be compared. Participants will be asked to evaluate the visual performance of each lens after 1 week of wear through a questionnaire.

Hypothesis: It is expected that one week's wear of the peripheral myopic defocus contact lens will cause an increase in blood vessel density and a thickening of the choroid compared with initial measurements. A decrease in blood vessel density and choroidal thinning is expected after one week's wear of the spherical soft lens (hyperopic defocus), compared with baseline. Both lenses will be well tolerated during daily activities.

ELIGIBILITY:
Inclusion Criteria:

* · Astigmatism ≤ 1.00 D

  * Myopia between -0.50 and -4.00D
  * Aged between 18 and 35
  * Binocular acuity of 6/6 or better

Exclusion Criteria:

* · Recent intake (< 3 months) of medication affecting blood pressure (e.g. hypotensive, anovulant, CNS stimulant, etc.).

  * Corneal dystrophy or irregularity
  * Use of topical ocular medications
  * Smoking (tobacco or marijuana)
  * Have contraindications to wearing soft contact lenses
  * Being currently under myopia control treatment or had been under control in the last 3 months
  * Being pregnant or breast-feeding
  * History of refractive surgery
  * Addiction to drugs or alcohol

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of Retinal blood vessel density measured by Triton OCT-A | Measurement done at baseline and after 1 week of contact lens wear
  The TRITON angiographic optical coherence tomograph will be used in this research project. OCT-A is a non-invasive angiography that enables changes in retinal vascularization to be observed. This is achieved by analyzing the movement of erythrocytes in blood vessels using a series of B-scans. Retinal vessel density will be measured at the macular area and at the optic nerve head. (2 scans)

OTHER OUTCOMES:
Evaluation of the choroidal thickness at the macular area | Measurement done at baseline and after 1 week of contact lens wear
  A 3D scan (OCT- Heidelberg) 6.0mm x 6.0mm will be performed for analysis of choroidal thickness in the different ETDRS quadrants. Choroidal thickness data per quadrant (1-5) will be available in the 6mm CSI analysis (BM-CSI)

CONTACTS AND LOCATIONS:
Overall Officials: Langis Michaud, OD MS, Principal Investigator — Universite de Montreal
Locations (1):
- Universite de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agawa T, Miura M, Ikuno Y, Makita S, Fabritius T, Iwasaki T, Goto H, Nishida K, Yasuno Y. Choroidal thickness measurement in healthy Japanese subjects by three-dimensional high-penetration optical coherence tomography. Graefes Arch Clin Exp Ophthalmol. 2011 Oct;249(10):1485-92. doi: 10.1007/s00417-011-1708-7. Epub 2011 May 10. PMID 21556938
- [Background] Harb E, Hyman L, Gwiazda J, Marsh-Tootle W, Zhang Q, Hou W, Norton TT, Weise K, Dirkes K, Zangwill LM; COMET Study Group. Choroidal Thickness Profiles in Myopic Eyes of Young Adults in the Correction of Myopia Evaluation Trial Cohort. Am J Ophthalmol. 2015 Jul;160(1):62-71.e2. doi: 10.1016/j.ajo.2015.04.018. Epub 2015 Apr 18. PMID 25896460
- [Background] Ostrin LA, Harb E, Nickla DL, Read SA, Alonso-Caneiro D, Schroedl F, Kaser-Eichberger A, Zhou X, Wildsoet CF. IMI-The Dynamic Choroid: New Insights, Challenges, and Potential Significance for Human Myopia. Invest Ophthalmol Vis Sci. 2023 May 1;64(6):4. doi: 10.1167/iovs.64.6.4. PMID 37126359
- [Background] Chiang ST, Phillips JR, Backhouse S. Effect of retinal image defocus on the thickness of the human choroid. Ophthalmic Physiol Opt. 2015 Jul;35(4):405-13. doi: 10.1111/opo.12218. Epub 2015 May 24. PMID 26010292
- [Background] Wang D, Chun RK, Liu M, Lee RP, Sun Y, Zhang T, Lam C, Liu Q, To CH. Optical Defocus Rapidly Changes Choroidal Thickness in Schoolchildren. PLoS One. 2016 Aug 18;11(8):e0161535. doi: 10.1371/journal.pone.0161535. eCollection 2016. PMID 27537606
- [Background] Breher K, Garcia Garcia M, Ohlendorf A, Wahl S. The effect of the optical design of multifocal contact lenses on choroidal thickness. PLoS One. 2018 Nov 16;13(11):e0207637. doi: 10.1371/journal.pone.0207637. eCollection 2018. PMID 30444900
- [Background] Campbell JP, Zhang M, Hwang TS, Bailey ST, Wilson DJ, Jia Y, Huang D. Detailed Vascular Anatomy of the Human Retina by Projection-Resolved Optical Coherence Tomography Angiography. Sci Rep. 2017 Feb 10;7:42201. doi: 10.1038/srep42201. PMID 28186181
- [Background] Swiatczak B, Schaeffel F, Calzetti G. Imposed positive defocus changes choroidal blood flow in young human subjects. Graefes Arch Clin Exp Ophthalmol. 2023 Jan;261(1):115-125. doi: 10.1007/s00417-022-05842-z. Epub 2022 Sep 29. PMID 36171460
- [Background] Wang E, Zhao X, Yang J, Chen Y. Visualization of deep choroidal vasculatures and measurement of choroidal vascular density: a swept-source optical coherence tomography angiography approach. BMC Ophthalmol. 2020 Aug 5;20(1):321. doi: 10.1186/s12886-020-01591-x. PMID 32758186
- Available data/document: Study Protocol — https://nagano.umontreal.ca/login — Protocol and other documentation available upon request to the principal investigator email

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT06527274/Prot_SAP_ICF_000.pdf